CLINICAL TRIAL: NCT00084344
Title: A Prospective, Randomized, Placebo-Controlled Trial of the Effects of 4-Hydroxytamoxifen Gel on Breast Density, Salivary Sex Steroids, and Quality of Life in Premenopausal Women
Brief Title: Effect of 4-Hydroxytamoxifen Gel on Breast Density, Salivary Sex Steroids, and Quality of Life in Premenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Screening
Other Study IDs: NCI 00B3; NU-NCI-00B3; NU-3; NU-0365-011
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — afimoxifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: 4-hydroxytamoxifen
Procedure: breast imaging study
Procedure: radiomammography

SUMMARY:
RATIONALE: High estrogen levels may be associated with dense breast tissue and an increased risk of developing breast cancer. 4-hydroxytamoxifen gel (a substance made when tamoxifen breaks down in the body) may be effective in reducing breast density by reducing estrogen levels with fewer side effects than tamoxifen. This may improve quality of life and the ability to detect breast cancer with screening mammography.

PURPOSE: Randomized screening study to determine the effect of 4-hydroxytamoxifen gel on breast density, salivary sex steroids (hormones), and quality of life in premenopausal women.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of 4-hydroxytamoxifen gel on breast density, as measured by digital mammography, in premenopausal women.
* Determine the effect of this gel on breast density in these participants, as defined by the BIRADS lexicon.

Secondary

* Determine the effect of this gel on salivary sex steroid levels in these participants.
* Determine the effect of this gel on quality of life of these participants.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Participants are randomized to 1 of 2 treatment arms.

* Arm I: Participants apply 4-hydroxytamoxifen gel in 4 metered doses daily to each breast beginning on the first day after cessation of the first menstrual period after digital mammography is performed.
* Arm II: Participants apply placebo gel as in arm I. In both arms, treatment continues for 1 year.

In both arms, participants collect daily saliva samples for 4 menstrual cycles during the study. Three of the saliva collections occur during the cycles encompassing the time periods when imaging studies are performed (months 0, 6, and 12). The fourth collection takes place during the first month that gel is applied to the breast.

Participants also undergo digital mammography at baseline, 6 months, and 1 year.

Participants who develop clinical breast problems considered suspicious for cancer discontinue study treatment until a histological diagnosis is established. Those found to have breast cancer are removed from the study and those with benign disease continue the study. If an excisional biopsy is performed, density measurements are made on the opposite breast.

Quality of life is assessed at baseline, 1 month, 6 months, and 1 year.

PROJECTED ACCRUAL: A total of 100 participants (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Premenopausal as determined by a menstrual history of no change in menstrual pattern within the past 6 months
* Undergoing mammography at least annually
* No prior breast cancer
* No clinical breast abnormalities suspicious for cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 30 to 50

Sex

* Female

Menopausal status

* See Disease Characteristics

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective barrier contraception
* No medical or psychiatric disorder that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 3 months since prior oral contraceptives or other estrogen- or progesterone-containing drugs
* No prior tamoxifen for more than 1 month duration
* No concurrent oral contraceptives or other estrogen- or progesterone-containing drugs
* No other concurrent antiestrogen medications

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2003-04; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seema A. Khan, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States